CLINICAL TRIAL: NCT03404362
Title: A Two-center Phase II, Non-randomized Study of MRgFUS Versus EBRT in Patients With Metastatic Non-spinal Bone Disease: Palliative Strategy for Cancer-Induced Bone Pain
Brief Title: MRgFUS Versus EBRT in Patients With Metastatic Non-spinal Bone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Alessandro Napoli, Associate Professor, University of Roma La Sapienza
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BM-Fus Vs RT
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Secondary Bone Cancer; Bone Metastases
Keywords: Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRgFUS (Active Comparator): The treatment process begins with the physician acquiring a set of MR images, identifying target volume(s) of tissue to ablate, and then drawing the treatment contours.
  The therapy planning software computes the type and number of sonications required to treat the defined region while minimizing total treatment time. MR images taken during the sonication provide a diagnostic quality image of the target tissue and a quantitative, real-time temperature map overlay to confirm the therapeutic effect of the treatment
  Interventions: Procedure: Bone Metastases Pain treatment
- EBRT (Active Comparator): Patient would undergo single fraction of external beam radiation to a dose of 8Gy or a session of 10 fractions of external beam radiations at 3Gy per fraction for two weeks.
  Interventions: Procedure: Bone Metastases Pain treatment

INTERVENTIONS:
Procedure: Bone Metastases Pain treatment — Comparative treatments to test if MRgFUS is an effective non-invasive and safe treatment for the palliation of metastatic bone tumors with a low incidence of co-morbidity as compared to EBRT (gold-standard)

SUMMARY:
The objective of this trial is to collect and compare safety and effectiveness data of Magnetic Resonance guided Focused Ultrasound (MRgFUS) using the ExAblate 2100 device and radiotherapy in the treatment of metastatic bone tumors.

This study is designed as a prospective, double arm, non-randomized study with External Beam radiation therapy (EBRT) serving as control arm.

The study hypothesis is that MRgFUS is an effective non-invasive and safe treatment for the palliation of metastatic bone tumors with a low incidence of co-morbidity as compared to EBRT.

DETAILED DESCRIPTION:
This is a prospective, phase II, open-label, non-randomized, double arm study to collect data on safety and effectiveness of ExAblate MRgFUS and EBRT treatments of metastatic bone tumors. Following treatment assignment and treatment itself, subjects will be followed for up for 12 months to evaluate pain relief as well as quality of life. Additional data regarding dosage and frequency of analgesic consumption for the management of the bone tumor induced pain will also be collected. MRI of the treated lesion will be obtained 3 and 6 months post therapy to evaluate effect on the lesion in both radiation and MRgFUS arms. This is clinically acceptable and widely utilized diagnostic method in follow up of this patient population.

Data will be collected for a total of 184 patients, 92 patients treated by EBRT and another 92 patients treated by FUS.

Treating physician, as of his/her normal practice, might offer additional treatment of other type in cases where pain score of the treated lesion will not improve by at least 2 points, and will remain 4 or greater. Additional treatment may be performed up to one month following treatment. Prior to offering alternative treatment, an MRI will be performed to evaluate effect on the lesion. Patient receiving another treatment, different from the initial one (i.e. patient initially treated with FUS is now treated by EBRT) will be considered as treatment failures for the primary analysis and their post-x-over follow-up results will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 years and older.
2. Able and willing to give consent and to attend all study visits
3. Patients with bone metastasis or primary bone lesion identifiable by imaging techniques.
4. Worst NRS Pain Score of ≥ 4 from the tumor to be treated.
5. Each targeted tumor is accessible to both ExAblate and EBRT (ExAblate accessible lesions are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5), please see ExAblate "Information for Prescribers".
6. Targeted tumor area is smaller than 100cm2.
7. Tumor clearly visible by non-contrast MRI.
8. No radiation therapy to selected lesion during one month prior to enrollment.
9. Radiation therapy to selected lesion is not contraindicated
10. Bisphosphonate, chemo or hormone therapy intake should remain stable throughout follow up duration.

Exclusion Criteria:

1. Patients who either need pre-treatment surgical stabilization of the affected bony structure
2. Targeted tumor is in a vertebra body or in the posterior aspects of the vertebral column other than Lumbar vertebra (L3 - L5) and Sacral vertebra (S1 - S5).
3. Targeted tumor is in the skull.
4. Patients on anti-coagulation therapy or with an underlying uncontrolled bleeding disorder.
5. Patients with life expectancy < 6-Months.
6. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication.
   * Patients with documented myocardial infarction within last 40 days to protocol entry.
   * Congestive heart failure NYHA Class IV
7. Severe hypertension (diastolic BP > 100 on medication).
8. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted ferromagnetic objects/devices.
9. Known intolerance or allergies to MRI contrast agent (e.g. Gadolinium or Magnevist)
10. KPS score of below 60
11. Severe cerebro-vascular disease (multiple CVA or CVA within 6 months)
12. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
13. Target tumor is less then 1cm from spinal cord, skin, or hollow viscera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Determine the effect of MRgFUS in terms of level of pain relief and decrease in analgesics/opiate and improved quality of life. | one month
  The key points that this study will capture are as follows:
  Capture patient-based pain assessment using a NRS pain scale of 0-10 with anchored points in conjunction with a body diagram, capturing worst and average pain score.
  Response rates were defined as follows:
  1. Complete response: NRS of 0 with no concomitant increase in analgesic intake (stable or reduced OMED);
  2. Partial response: a reduction in NRS ≥ 2 points from baseline without an analgesic increase or analgesic reduction ≥ 25% from baseline without an increase in pain;
  3. Pain progression: an increase in NRS ≥ 2 points above baseline with stable OMED or an increase ≥ 25% in OMED from baseline with NRS stable or 1 point above baseline;
  4. Indeterminate response: any response not captured by definitions 1, 2 and 3

OTHER OUTCOMES:
Brief Pain Inventory (BPI) | 12 months
  Brief Pain Inventory (BPI) will be used to capture patient estimates of their global rating of change in pain at the treatment site to anchor change scores on a given instrument. Clinically significant responses were defined as a reduction ≥ 2 from baseline
Quality of Life Questionnaire Cancer 15 Palliative Care (QLQ-C15-PAL) | 12 months
  QLQ-C15-PAL will be used to capture patient estimates of their global rating of change in pain at the treatment site to anchor change scores on a given instrument. Clinically significant responses were defined as a reduction ≥5 points from baseline
Quality of Life Questionnaire Bone Metastases 22 (QLQ-BM22) | 12 months
  QLQ-C15-PAL will be used to capture patient estimates of their global rating of change in pain at the treatment site to anchor change scores on a given instrument. Clinically significant responses were defined as a reduction ≥8 points from baseline
Compare incidence and severity of adverse events associated with the ExAblate MRgFUS bone system to that of EBRT. | 12 months
  Safety of both treatments will be determined by an evaluation of the incidence and severity of device and procedure related complications from the first / treatment day visit through the 12-Months post-treatment time point. Adverse events were categorized according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Alessandro Napoli, Rome
  - Sapienza University of Rome, Policlinico Umberto I Hospital, Rome

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anzidei M, Napoli A, Sacconi B, Boni F, Noce V, Di Martino M, Saba L, Catalano C. Magnetic resonance-guided focused ultrasound for the treatment of painful bone metastases: role of apparent diffusion coefficient (ADC) and dynamic contrast enhanced (DCE) MRI in the assessment of clinical outcome. Radiol Med. 2016 Dec;121(12):905-915. doi: 10.1007/s11547-016-0675-9. Epub 2016 Aug 27. PMID 27567615
- [Background] Huisman M, ter Haar G, Napoli A, Hananel A, Ghanouni P, Lovey G, Nijenhuis RJ, van den Bosch MA, Rieke V, Majumdar S, Marchetti L, Pfeffer RM, Hurwitz MD. International consensus on use of focused ultrasound for painful bone metastases: Current status and future directions. Int J Hyperthermia. 2015 May;31(3):251-9. doi: 10.3109/02656736.2014.995237. Epub 2015 Feb 13. PMID 25677840
- [Background] Hurwitz MD, Ghanouni P, Kanaev SV, Iozeffi D, Gianfelice D, Fennessy FM, Kuten A, Meyer JE, LeBlang SD, Roberts A, Choi J, Larner JM, Napoli A, Turkevich VG, Inbar Y, Tempany CM, Pfeffer RM. Magnetic resonance-guided focused ultrasound for patients with painful bone metastases: phase III trial results. J Natl Cancer Inst. 2014 Apr 23;106(5):dju082. doi: 10.1093/jnci/dju082. PMID 24760791
- [Background] Napoli A, Anzidei M, Marincola BC, Brachetti G, Noce V, Boni F, Bertaccini L, Passariello R, Catalano C. MR imaging-guided focused ultrasound for treatment of bone metastasis. Radiographics. 2013 Oct;33(6):1555-68. doi: 10.1148/rg.336125162. PMID 24108551
- [Background] Napoli A, Anzidei M, Marincola BC, Brachetti G, Ciolina F, Cartocci G, Marsecano C, Zaccagna F, Marchetti L, Cortesi E, Catalano C. Primary pain palliation and local tumor control in bone metastases treated with magnetic resonance-guided focused ultrasound. Invest Radiol. 2013 Jun;48(6):351-8. doi: 10.1097/RLI.0b013e318285bbab. PMID 23571832